CLINICAL TRIAL: NCT03852160
Title: A Randomized, Double-Blind, Active-Controlled, International, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Flexibly-dosed Esketamine Nasal Spray Plus a New Standard-of-care Oral Antidepressant or Placebo Nasal Spray Plus a New Standard-of-care Oral Antidepressant in Adult and Elderly Participants With Treatment-resistant Depression
Brief Title: A Study of Esketamine Nasal Spray Plus a New Standard-of-care Oral Antidepressant or Placebo Nasal Spray Plus a New Standard-of-care Oral Antidepressant in Adult and Elderly Participants With Treatment-resistant Depression
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: New design was developed to better fit company strategy, a new study has replaced 5413541TRD3011 study
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108567; 2018-001890-26 (EudraCT Number); 54135419TRD3011 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2019-02-12; First posted 2019-02-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Esketamine; Escitalopram; Sertraline; Duloxetine Hydrochloride; Mirtazapine; agomelatine; Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Esketamine + Oral Antidepressants (Experimental): Participants will receive esketamine as nasal spray (28 milligram [mg] [initial dose for elderly participants 65-74 years of age] on Day 1 and then uptitrated to 56 mg on Day 4, 56 mg [initial dose for adult participants aged 18-64 years and may be used for all age groups throughout the study] or 84 mg [maximum uptitrated esketamine dose]) twice-weekly with a flexible dose regimen from Day 1 until Day 28 (Week 4), once weekly from Week 5 to Week 8 and once-weekly or once every other week from Week 9 to Week 32. The dose may be increased/decreased at any visit or may remain the same as determined by the investigator based on efficacy and tolerability. In addition, participants will initiate a new standard-of-care oral anti depressants (AD) (escitalopram, sertraline, duloxetine, agomelatine, mirtazapine, bupropion or trazodone prolonged release) on Day 1, taken daily for the duration of the study.
  Interventions: Drug: Esketamine 28 mg; Drug: Esketamine 56 mg; Drug: Esketamine 84 mg; Drug: Escitalopram; Drug: Sertraline; Drug: Duloxetine; Drug: Mirtazapine; Drug: Agomelatine; Drug: Bupropion; Drug: Trazodone Prolonged Release
- Placebo + Oral Antidepressants (Active Comparator): Participants will receive matching placebo as nasal spray twice-weekly with a flexible dose regimen from Day 1 until Day 28 (Week 4), once weekly from Week 5 to Week 8 and once-weekly or once every other week from Week 9 to Week 32. The dose may be increased/decreased at any visit or may remain the same as determined by the investigator based on efficacy and tolerability. In addition, participants will initiate a new standard-of-care oral AD (escitalopram, sertraline, duloxetine, agomelatine, mirtazapine, bupropion or trazodone prolonged release) on Day 1, taken daily for the duration of the study.
  Interventions: Drug: Placebo; Drug: Escitalopram; Drug: Sertraline; Drug: Duloxetine; Drug: Mirtazapine; Drug: Agomelatine; Drug: Bupropion; Drug: Trazodone Prolonged Release

INTERVENTIONS:
Drug: Esketamine 28 mg — Participants will receive 28 mg esketamine as nasal spray (Initial dose for elderly participants with 65-74 years of age on Day 1 and then uptitrated to 56 mg on Day 4).
  Other Names: JNJ-54135419
  Arms: Esketamine + Oral Antidepressants
Drug: Esketamine 56 mg — Participants will receive 56 mg esketamine as nasal spray (Initial dose for participants with 18-64 years of age) on Day 1. The dose may be increased/may remain same based on the efficacy and tolerability. Participants with 65 to 74 years of age will receive esketamine 56 mg from Day 4 onwards.
  Other Names: JNJ-54135419
  Arms: Esketamine + Oral Antidepressants
Drug: Esketamine 84 mg — Participants may receive 84 mg (maximum uptitrated esketamine dose). The dose may be decreased/may remain same based on the efficacy and tolerability.
  Other Names: JNJ-54135419
  Arms: Esketamine + Oral Antidepressants
Drug: Placebo — Participants will receive matching placebo as nasal spray.
  Arms: Placebo + Oral Antidepressants
Drug: Escitalopram — Escitalopram can be selected as the oral antidepressant medication based on investigator's discretion. The initial dose for escitalopram is 5 mg once daily (for elderly participants) and 10 mg once daily (for adults). The dose may be increased to 10 mg (for elderly participants) and 20 mg (for adults) once daily at the discretion of treating physician/investigator.
Drug: Sertraline — Sertraline can be selected as the oral antidepressant medication based on investigator's discretion. The initial dose for sertraline is 50 mg once daily and may be increased up to 200 mg once daily.
Drug: Duloxetine — Duloxetine can be selected as the oral antidepressant medication based on investigator's discretion. The initial dose for duloxetine is 60 mg once daily and may be increased to 120 mg once daily.
Drug: Mirtazapine — Mirtazapine can be selected as the oral antidepressant medication based on investigator's discretion. The initial dose for mirtazapine is 15 to 30 mg once daily and may be increased to 45 mg once daily.
Drug: Agomelatine — Agomelatine can be selected as the oral antidepressant medication based on investigator's discretion. The initial dose for agomelatine is 25 mg once daily and may be increased to 50 mg once daily after 2 weeks.
Drug: Bupropion — Bupropion can be selected as the oral antidepressant medication based on investigator's discretion. The initial dose for bupropion is 150 mg once daily and may be increased to 300 mg once daily after 4 weeks.
Drug: Trazodone Prolonged Release — Trazodone prolonged release can be selected as the oral antidepressant medication based on investigator's discretion. The initial dose for trazodone prolonged release is 75 to 150 mg once or twice daily and may be increased up to 450 mg (adults) and 300 mg (elderly).

SUMMARY:
The purpose of this study is to evaluate the efficacy of treating participants with treatment-resistant depression (TRD) who have failed at least 2 (and no more than 6) prior antidepressant (AD) treatments in the current moderate to severe depressive episode with flexibly-dosed esketamine nasal spray plus a newly initiated oral standard-of-care AD compared with placebo nasal spray plus a newly-initiated standard-of-care oral AD, in achieving remission and staying relapse-free after remission.

DETAILED DESCRIPTION:
Depression is a major cause of morbidity and mortality, with global estimates of 300 million treated and untreated individuals worldwide. In its severe forms, depression is the most common diagnosis associated with suicide. Esketamine (S-ketamine) is the S-enantiomer of ketamine. Ketamine profoundly affects fast excitatory glutamate transmission, increases brain-derived neurotrophic factor release, and stimulates synaptogenesis, in contrast to conventional antidepressants (ADs) which are modulatory transmitters. The goal of any new antidepressant (AD) treatment would be the rapid and long-lasting relief of depressive symptoms. The study includes screening phase (2 weeks, with possible extension up to 4 weeks), Induction phase (Week 1 to Week 4), Maintenance once-weekly phase (Week 5 to Week 8), Maintenance flexible-frequency phase (Week 9 to Week 32) and Follow-up phase (2 Weeks Duration). Total duration of study will be approximately up to 36 weeks. The safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* At screening, each participant must meet Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) diagnostic criteria for single episode major depressive disorder (MDD) or recurrent MDD, without psychotic features, based on clinical assessment and confirmed by the Mini International Neuropsychiatric Interview (MINI)
* At baseline, each participant must have an Inventory of Depressive Symptomology Clinician-Rated 30 Items Scale (IDS-C30) total score of greater than or equal to (>= ) 34
* At screening, participants must have had a documented nonresponse to at least 2 but not more than 6 oral antidepressants (AD) treatments taken at adequate dosage and for adequate duration within the current episode of depression evaluated retrospectively. Nonresponse documentation at screening must include the sequence of retrospectively failed antidepressants and combination and or augmentation for retrospectively failed antidepressants
* Must be medically stable based on physical examination, medical history, vital signs (including blood pressure). If there are any abnormalities that are not specified in the inclusion and exclusion criteria, their clinical significance must be determined by the investigator and recorded in the participant's source documents
* Must be comfortable with self-administration of nasal medication and be able to follow the nasal administration instructions provided
* A woman of childbearing potential must have a negative highly sensitive serum (Beta human chorionic gonadotropin [Beta hCG]) at screening and a negative urine pregnancy test prior to the first dose of study intervention on Day 1 of the induction phase prior to randomization

Exclusion Criteria:

* Depressive symptoms that have previously not responded to any of the following:

a Esketamine or ketamine in a major depressive episode per clinical judgment, or b All of the classes of oral ADs in the study or an adequate AD augmentation/combination therapy in the current major depressive episode, or c An adequate course of treatment with electroconvulsive therapy in the current major depressive episode, defined as at least 7 treatments with unilateral/bilateral electroconvulsive therapy

* Received vagal nerve stimulation (VNS) or has received deep brain stimulation (DBS) in the current episode of depression
* Has a current or prior DSM-5 diagnosis of a psychotic disorder or MDD with psychotic features, bipolar or related disorders (confirmed by the MINI), intellectual disability, autism spectrum disorder, borderline personality disorder, antisocial personality disorder
* Has homicidal ideation or intent, per the investigator's clinical judgment; or has suicidal ideation with some intent to act within 1 month prior to screening, per the investigator's clinical judgment; or based on the Columbia Suicide Severity Rating Scale (C-SSRS), corresponding to a response of "Yes" on Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) for suicidal ideation on the C SSRS, or a history of suicidal behavior within the past year prior to screening. Participants reporting suicidal ideation with intent to act or suicidal behavior prior to the start of the induction phase should also be excluded
* History of moderate or severe substance use disorder or severe alcohol use disorder according to DSM-5 criteria, except nicotine or caffeine, within 6 months before the start of the screening or current clinical signs
* Has other inflammatory diseases that might confound the evaluations of benefit of guselkumab therapy, including but not limited to Rheumatoid arthritis (RA), axial spondyloarthritis (this does not include a primary diagnosis of psoriatic spondylitis [PsA] with spondylitis), systemic lupus erythematosus, or Lyme disease

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2021-07-25 (Estimated); Study Completion 2021-07-25 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Remission as Assessed by the Montgomery-Asberg Depression Rating Scale (MADRS) (Total Score of less than or Equal to [<=] 10) at the end of Week 8 | Week 8
  Percentage of participants with remission as assessed by the MADRS (total score of <= 10) will be reported and compared between treatment arms. The MADRS is a clinician-rated scale designed to measure depression severity. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms).These item scores are summed up to yield a total score. The range of the total score is 0 to 60. Higher scores represent a more severe condition. The MADRS evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, inability to feel (interest level), pessimistic thoughts, and suicidal thoughts.

SECONDARY OUTCOMES:
Percentage of Participants with Remission at Week 8 Without Relapse Until Week 32 | Week 32
  Percentage of participants with remission (as assessed by MADRS [total score of <= 10) at Week 8 without relapse until Week 32 will be reported at Week 32. A relapse is defined any of following- a) Worsening of depressive symptoms in participants who have achieved remission, as indicated by MADRS total score greater than equal to (>=) 22 confirmed by one additional assessment of MADRS total score >= 22 within next 5 to 15 days (until Week 32). Date of second MADRS assessment will be used for date of relapse; b) Any psychiatric hospitalization for worsening of depression, hospitalization for suicide prevention or completed suicide. For any of these events, start date of hospitalization will be used for date of relapse, c) Suicide attempt or any other clinically relevant event determined per the investigator's clinical judgment to be indicative of a relapse of depressive illness, but for which participant was not hospitalized. The onset of event will be used for date of relapse.
Change from Baseline in Clinician-reported MADRS Scale Score | Baseline, up to 32 Week
  The MADRS is a clinician-rated scale designed to measure depression severity. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms). These item scores are summed up to yield a total score. The range of the total score is 0 to 60. Higher scores represent a more severe condition. The MADRS evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, inability to feel (interest level), pessimistic thoughts, and suicidal thoughts.
Change in MADRS Total Score from Baseline at Week 4 | Baseline, Week 4
  The MADRS is a clinician-rated scale designed to measure depression severity. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms). These item scores are summed up to yield a total score. The range of the total score is 0 to 60. Higher scores represent a more severe condition. The MADRS evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, inability to feel (interest level), pessimistic thoughts, and suicidal thoughts.
Change from Baseline in Patient Health Questionnaire (PHQ) 9-item Total Score | Baseline, up to 32 Weeks
  The PHQ-9 is a 9-item, patient-reported outcome (PRO) measure to assess depressive symptoms. The scale scores each of the 9-symptom domains of the Diagnostic and Statistical Manual of Mental Disorders, fifth edition major depressive disorder (DSM-5 MDD) criteria. Each item is rated on a 4 point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms.
Change from Baseline in Clinical Global Impression - Severity (CGI-S) Scale Score | Baseline, up to 32 Weeks
  The CGI-S rating scale is a global assessment that measures the clinician's impression of the severity of illness of the participant. A rating scale of 1 to 7 is used, with 1="normal, not at all ill" and 7="among the most extremely ill".
Clinical Global Impression - Change (CGI-C) Scale Score | Up to 32 Weeks
  The CGI-C rating scale is a global assessment that measures the clinician's impression illness change. CGI-C scores range from 1 (very much improved) through to 7 (very much worse).
Change from Baseline in Sheehan Disability Scale (SDS) Total Score | Baseline, up to 32 Weeks
  The SDS, a patient-reported outcome measure, is a 5-item questionnaire that has been widely used and accepted for assessment of functional impairment and associated disability. The first 3 items cover (1) work/school, (2) social life, and (3) family life/home responsibilities using a rating scale from 0 to 10. The score for the first 3 items are summed to create a total score of 0 to 30, where higher score indicates greater impairment.
Change from Baseline in Health-Related Quality of life Status as Assessed by 36-item Short-Form Health Survey (SF-36) Domain Scores | Baseline, up to 32 Weeks
  The Short-Form-36 (SF-36) is a 36-item questionnaire which measures quality of life (QoL) across 8 domains, which are both physically and emotionally based. The 8 domains that the SF36 measures are as follows: physical functioning; role limitations due to physical health; role limitations due to emotional problems; energy/fatigue; emotional wellbeing; social functioning; pain; general health. For each of the 8 domains that the SF-36 measures, an aggregate score is produced. The scores range from 0 (lowest or worst possible level of functioning) to 100 (highest or best possible level of functioning).
Change from Baseline in Quality of Life in Depression Scale (QLDS) Total Score | Baseline, up to 32 Weeks
  The QLDS is a disease specific PRO designed to assess health related quality of life in patients with Major Depressive Disorder. The instrument has a recall period of "at the moment", contains 34-items with "yes"/"no" response options and takes approximately 5-10 minutes to complete. The total score is computed as sum of the items with range from 0 (good quality of life) to 34 (very poor quality of life).
Change from Baseline in European Quality of Life (EuroQol) Group, 5 Dimension, 5-Level (EQ-5D-5L): EQ-VAS | Baseline, up to 32 weeks
  The EQ-5D-5L is standardized instrument for use as measure of health outcome, primarily designed for self-completion by respondents. It consists of EQ-5D-5L descriptive system and EQ-VAS. The EQ-VAS rating "health today" with range from 0 (worst imaginable health state) to 100 (best imaginable health state).
Change from Baseline in European Quality of Life (EuroQol) Group, 5 Dimension, 5-Level (EQ-5D-5L): Health Status Index | Baseline, up to 32 Weeks
  The EQ-5D-5L is standardized instrument for use as measure of health outcome, primarily designed for self-completion by respondents. It consists of EQ-5D-5L descriptive system and EQ-VAS. EQ-5D-5L descriptive system comprises the following 5 dimensions: Mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of 5 dimensions is divided into 5 levels of perceived problems (1 indicating no problem, 2 indicating slight problems, 3 indicating moderate problems, 4 indicating severe problems, 5 indicating extreme problems). Participant selects an answer for each of 5 dimensions considering the response that best matches his or her health "today". The responses to the 5 dimensions are used to compute a single score ranging from zero (0.0- worst health state) to 1 (1.0- better health state) representing the general health status of the individual.
Change from Baseline in Work Productivity and Activity Impairment- Specific Health Problem (WPAI-SHP) Questionnaire Scores | Baseline, up to 32 Weeks
  WPAI-SHP is a validated short instrument that assesses impairment in work and other regular activities over the past 7 days. WPAI produces four types of scores: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment. The WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, that is, worse outcomes.
Medical Resource Utilization | Up to 32 weeks
  Number of medical care encounters and treatments (including physician or emergency room visits, tests and procedures, and medications, and other procedures) will be reported.
Number of Participants with Treatment-Emergent Adverse Events | Up to 32 Weeks
  An adverse event (AE) is any untoward medical occurrence attributed to study drug in a participant who received study drug.
Suicidal ideation and behavior as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) Score | Baseline, up to 32 weeks
  Suicidal ideation or behavior will be measured using C-SSRS score. C-SSRS is a clinician rated assessment of suicidal behavior and/ or intent. Scale consists of 28 items in 4 sections: suicide behavior, actual attempts, suicidal ideation, and intensity of ideation. Suicidal ideation consists of 5 yes/no items: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intention to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent. Worsening of suicidal ideation will be an increase in severity of suicidal ideation from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency